CLINICAL TRIAL: NCT05400421
Title: Validation of Photoplethysmography Device for the Measurement of Aortic Pulse Wave Velocity Against Carotid-Femoral Values From Piezoelectric Sensors
Brief Title: Validation of Optical Device for Aortic Pulse Wave Velocity Measurement
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: VitalSines International Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: OBA-MAPWV
Record Dates: First submitted 2022-05-27; First posted 2022-06-01 (Actual); Last update posted 2022-06-06 (Actual); Status verified 2022-06

CONDITIONS: Aortic Pulse Wave Velocity
Keywords: aortic pulse wave velocity; plethysmography
MeSH Terms: interventions — Drug Delivery Systems; Methods; Blood Pressure

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Device Calibration & Algorithm Training: The data obtained from this group will be used to a) quantify the relationship between PWV measured at the groin versus the thigh for less intrusive future piezo sensor placement and b) train the proposed device for the next cohort.
  Interventions: Device: System & Method for Monitoring Aortic Pulse Wave Velocity & Blood Pressure
- Device & Algorithm Testing: The gold-standard and new device values will be collected from this group to validate the previously trained system.
  Interventions: Device: System & Method for Monitoring Aortic Pulse Wave Velocity & Blood Pressure

INTERVENTIONS:
Device: System & Method for Monitoring Aortic Pulse Wave Velocity & Blood Pressure — Carotid-femoral aortic pulse wave velocity will be compared against values collected from the oximeter system. The former is assessed by placing piezoelectric pressure sensors at three locations: the right common carotid artery, the right common femoral artery (groin), and the right superficial femoral artery (thigh). The oximeter will be secured on the right index finger. Simultaneous data collection will occur for both methods, with each trail lasting 60 seconds.

SUMMARY:
Existing techniques available for capturing reliable aortic pulse wave velocity measurements and estimating aortic stiffness are costly and require technical expertise. The purpose of this research is to investigate an oximeter device performance as a stand-alone aortic pulse wave velocity (PWV) measurement instrument. By validating this device and its measurements against the gold-standard method of carotid-femoral readings, we aim to demonstrate that the proposed method is an comparably effective in terms of the metrics (Mean difference, standard deviation, correlation, etc.) outlined by the Artery Society Guidelines.

ELIGIBILITY:
Inclusion Criteria:

-

Exclusion Criteria:

* History of cardiovascular disease
* Not in sinus rhythm/arrhythmia
* Pacemaker
* Impalpable arterial pulse
* Use of blood pressure medication
* Systolic blood pressure > 140
* Use of vasoactive medication
* Use of cholesterol medication
* Diabetes diagnosis
* Smokers
* BMI > 30 kg/m2
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Primary care clinic patients with a health cardiovascular background.
Sampling Method: Non-Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2022-06 (Estimated); Primary Completion 2022-07 (Estimated); Study Completion 2022-07 (Estimated)

PRIMARY OUTCOMES:
Aortic Pulse Wave Velocity | 6 measurements per subject, each lasting 60 seconds
  The speed at which a single pulse/heart beat propagates down the aorta.

CONTACTS AND LOCATIONS:
Overall Officials: Jess Goodman, M.D., Principal Investigator — VitalSines International Inc.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Safar ME, Levy BI, Struijker-Boudier H. Current perspectives on arterial stiffness and pulse pressure in hypertension and cardiovascular diseases. Circulation. 2003 Jun 10;107(22):2864-9. doi: 10.1161/01.CIR.0000069826.36125.B4. No abstract available. PMID 12796414
- [Background] Laurent S, Katsahian S, Fassot C, Tropeano AI, Gautier I, Laloux B, Boutouyrie P. Aortic stiffness is an independent predictor of fatal stroke in essential hypertension. Stroke. 2003 May;34(5):1203-6. doi: 10.1161/01.STR.0000065428.03209.64. Epub 2003 Apr 3. PMID 12677025
- [Background] Van Bortel LM, Laurent S, Boutouyrie P, Chowienczyk P, Cruickshank JK, De Backer T, Filipovsky J, Huybrechts S, Mattace-Raso FU, Protogerou AD, Schillaci G, Segers P, Vermeersch S, Weber T; Artery Society; European Society of Hypertension Working Group on Vascular Structure and Function; European Network for Noninvasive Investigation of Large Arteries. Expert consensus document on the measurement of aortic stiffness in daily practice using carotid-femoral pulse wave velocity. J Hypertens. 2012 Mar;30(3):445-8. doi: 10.1097/HJH.0b013e32834fa8b0. PMID 22278144
- [Background] Xu SK, Hong XF, Cheng YB, Liu CY, Li Y, Yin B, Wang JG. Validation of a Piezoelectric Sensor Array-Based Device for Measurement of Carotid-Femoral Pulse Wave Velocity: The Philips Prototype. Pulse (Basel). 2018 Mar;5(1-4):161-168. doi: 10.1159/000486317. Epub 2018 Feb 8. PMID 29761092
- [Background] Kelly R, Hayward C, Avolio A, O'Rourke M. Noninvasive determination of age-related changes in the human arterial pulse. Circulation. 1989 Dec;80(6):1652-9. doi: 10.1161/01.cir.80.6.1652. PMID 2598428
- [Background] Chirinos JA, Segers P, Duprez DA, Brumback L, Bluemke DA, Zamani P, Kronmal R, Vaidya D, Ouyang P, Townsend RR, Jacobs DR Jr. Late systolic central hypertension as a predictor of incident heart failure: the Multi-ethnic Study of Atherosclerosis. J Am Heart Assoc. 2015 Mar 3;4(3):e001335. doi: 10.1161/JAHA.114.001335. PMID 25736440
- [Background] Ding FH, Fan WX, Zhang RY, Zhang Q, Li Y, Wang JG. Validation of the noninvasive assessment of central blood pressure by the SphygmoCor and Omron devices against the invasive catheter measurement. Am J Hypertens. 2011 Dec;24(12):1306-11. doi: 10.1038/ajh.2011.145. Epub 2011 Oct 6. PMID 21976274
- [Background] Pereira T, Maldonado J, Coutinho R, Cardoso E, Laranjeiro M, Andrade I, Conde J. Invasive validation of the Complior Analyse in the assessment of central artery pressure curves: a methodological study. Blood Press Monit. 2014 Oct;19(5):280-7. doi: 10.1097/MBP.0000000000000058. PMID 24892879
- [Background] Wang TW, Lin SF. Wearable Piezoelectric-Based System for Continuous Beat-to-Beat Blood Pressure Measurement. Sensors (Basel). 2020 Feb 5;20(3):851. doi: 10.3390/s20030851. PMID 32033495
- [Background] Park J, Seok HS, Kim SS, Shin H. Photoplethysmogram Analysis and Applications: An Integrative Review. Front Physiol. 2022 Mar 1;12:808451. doi: 10.3389/fphys.2021.808451. eCollection 2021. PMID 35300400
- [Background] I.B. Wilkinson, C.M. McEniery, G. Schillaci, P. Boutouyrie, P. Segers, A. Donald, et al. ARTERY Society guidelines for validation of non-invasive haemodynamic measurement devices: part 1, arterial pulse wave velocity Artery Res, 4 (2) (2010), p. 34